CLINICAL TRIAL: NCT04976504
Title: Early Warning for Desaturation by Oxygen Reserve Index During Induction of General Anesthesia
Brief Title: Early Warning for Desaturation by Oxygen Reserve Index
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019-06-1-018CC
Record Dates: First submitted 2021-07-07; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Desaturation of Blood; Anesthesia
Keywords: Oxygen reserve index; Induction of general anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Oxygen reserve index: Male and female patients aged 18 to 80 years with ASA physical status I to III scheduled for elective surgery with planned arterial catheter placement before induction of general anesthesia and did not match the exclusion criteria.
  Interventions: Device: Oxygen reserve index

INTERVENTIONS:
Device: Oxygen reserve index — This is an observational study of the routine clinical practice with no specific additional interventions required. The investigators enrolled the ASA physical status I to III patients scheduled for elective surgery with planned arterial catheter placement before induction. ORi and standard monitors were placed. The patients were preoxygenated and received anesthesia induction as routine clinical practice. Intubation was done by video-laryngoscope. The endotracheal tube was not connected to the breathing circuit to avoid apneic oxygenation. Ventilation was resumed when SpO2 fell to 90%. ORi and SpO2 were recorded every ten seconds.

SUMMARY:
During the induction of general anesthesia, the anesthesiologist needs to provide the oxygen supply to meet the patient's needs continuously. In the clinical scenario, the pulse oximeter is used as a standard to monitor hemoglobin oxygen saturation (SpO2) but is limited to assess the oxygenation status beyond the measurement of 100%. The Oxygen Reserve Index (ORi) is a dimensionless parameter between 0 and 1 that is related to real-time oxygenation reserve status. This study was designed to evaluate the duration of warning time for desaturation provided by different ORi alarm triggers during prolonged apnea in surgical patients. The primary endpoint was the duration of additional warning time provided by the ORi trigger. The secondary endpoint was the correlation of ORi and PaO2.

DETAILED DESCRIPTION:
This is an observational study of the routine clinical practice with no specific additional interventions required.

The investigators enrolled the American Society of Anesthesiologists (ASA) physical status I to III patients scheduled for elective surgery with planned arterial catheter placement before induction. Patients were positioned supine on the operating room table. Standard monitors and the ORi sensor were placed. The patients were preoxygenated with a facemask (flow rate of 8 to 10 liters/minute) for 3 minutes with spontaneous ventilation. Propofol (2-2.5 mg/kg), fentanyl (2-3 mcg/kg) and rocuronium (0.6-0.9 mg/kg) were administrated to achieve anesthesia induction during following 3 minutes. The patient was keeping ventilated manually by the anesthesiologist during the induction phase and intubated under direct visualization with a video-assisted laryngoscope at 6 minutes. The endotracheal tube was not connected to the breathing circuit to avoid apneic oxygenation. The patients remained apneic. Ventilation was resumed when SpO2 fell to 90%. ORi and SpO2 were recorded every ten seconds. Arterial blood is sampled every minute, from preoxygenation to resumed ventilation, to observe blood oxygen concentration changes.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 to 80 years with ASA physical status I to III scheduled for elective surgery with planned arterial catheter placement before induction of general anesthesia.

Exclusion Criteria:

* Age <18 years
* Inability to give primary consent
* Pregnancy
* History of chronic obstructive pulmonary disease (COPD)
* History of asthma
* Suspected difficult intubation
* Preoperative hemoglobin less than 10 mg/dl.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female patients aged 18 to 80 years with ASA physical status I to III scheduled for elective surgery with planned arterial catheter placement before induction of general anesthesia and did not match the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Additional warning time provided by ORi trigger | From time of starting preoxygenation until the time of SpO2 90%, assessed up to 20 minutes
  The ORi peak warning time was defined as the duration from ORi decreased by 0.05 from the plateau or peak values until SpO2 decreased to 90%. The ORi 0.55 warning time was defined as the duration from the ORi value was 0.55 to SpO2 90%. The SpO2 waring time was defined as the duration from SpO2 98% to 90%. The added warning time provided by ORi peak or ORi 0.55 was defined as the difference between ORi peak warning time, ORi 0.55 warning time, and SpO2 warning time. The investigators will check the duration of the additional warning time provided by the ORi trigger.

SECONDARY OUTCOMES:
Correlation between ORi and PaO2 | From time of starting preoxygenation until the time of SpO2 90%, assessed up to 20 minutes
  The Oxygen Reserve Index is a dimensionless parameter between 0 and 1 that is related to real-time oxygenation reserve status in the moderate hyperoxic range (PaO2 of about 100 to 200 mmHg). The investigators will check the correlation between ORi and PaO2 in our study.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Wei Cheng, MD, Principal Investigator — Taipei Veteran General Hospital, Taiwan
Locations (1):
- Department of Anesthesiology, Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Applegate RL 2nd, Dorotta IL, Wells B, Juma D, Applegate PM. The Relationship Between Oxygen Reserve Index and Arterial Partial Pressure of Oxygen During Surgery. Anesth Analg. 2016 Sep;123(3):626-33. doi: 10.1213/ANE.0000000000001262. PMID 27007078
- [Background] Scheeren TWL, Belda FJ, Perel A. The oxygen reserve index (ORI): a new tool to monitor oxygen therapy. J Clin Monit Comput. 2018 Jun;32(3):379-389. doi: 10.1007/s10877-017-0049-4. Epub 2017 Aug 8. PMID 28791567
- [Background] Szmuk P, Steiner JW, Olomu PN, Ploski RP, Sessler DI, Ezri T. Oxygen Reserve Index: A Novel Noninvasive Measure of Oxygen Reserve--A Pilot Study. Anesthesiology. 2016 Apr;124(4):779-84. doi: 10.1097/ALN.0000000000001009. PMID 26978143
- [Background] Fleming NW, Singh A, Lee L, Applegate RL 2nd. Oxygen Reserve Index: Utility as an Early Warning for Desaturation in High-Risk Surgical Patients. Anesth Analg. 2021 Mar 1;132(3):770-776. doi: 10.1213/ANE.0000000000005109. PMID 32815872
- [Derived] Cheng HW, Yeh CY, Chang MY, Ting CK, Chang PL. How early warning with the Oxygen Reserve Index (ORi) can improve the detection of desaturation during induction of general anesthesia? J Clin Monit Comput. 2022 Oct;36(5):1379-1385. doi: 10.1007/s10877-021-00776-z. Epub 2021 Dec 25. PMID 34953137